CLINICAL TRIAL: NCT05284344
Title: The Impact of Glucotoxicity on Gastric Emptying in Chinese Patients With Newly Diagnosed Type 2 Diabetes
Status: Completed | Type: Observational
Sponsor: University of Adelaide (Other)
Collaborators: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Tongzhi Wu, Principal Investigator, University of Adelaide
Other Study IDs: KY20220214-08
Record Dates: First submitted 2022-02-24; First posted 2022-03-17 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; gastric emptying; gut hormones; blood glucose; bile acid; glycaemia variability
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Hypoglycemic Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- patients with newly diagnosed type 2 diabetes: Newly diagnosed, drug-naïve, Chinese patients with type 2 diabetes.
  Interventions: Drug: Anti-Diabetics
- Non-diabetic control subjects

INTERVENTIONS:
Drug: Anti-Diabetics — The anti-diabetic treatments include insulin glargine, insulin aspart, GLP-1 receptor agonist, DPP-4 inhibitor, SGLT-2 inhibitor, metformin, sulfonylureas and/or gliclazide. Therapeutic dose of each drug follows recommendation by the treating doctor.
  Groups: patients with newly diagnosed type 2 diabetes

SUMMARY:
Gastric emptying is now recognized as a major determinant of the blood glucose response to carbohydrate in both health and type 2 diabetes (T2D). While patients with longstanding diabetes exhibit a high prevalence of delayed gastric emptying, i.e. gastroparesis, patients with fewer complications are often associated with accelerated gastric emptying, which exacerbates postprandial glycaemic excursions. Moreover, gastric emptying appears to be more rapid in Han Chinese patients with T2D, as compared to Caucasian patients with T2D.

The proposed study will (i) compare the rate of gastric emptying in newly diagnosed, Chinese patients with T2D to non-diabetic controls, (ii) evaluate the relationship between gastric emptying and glycaemic indices, including measures of glucose variability, and (iii) determine whether gastric emptying is altered by glucose-lowering therapies.

DETAILED DESCRIPTION:
A total of 100 newly diagnosed Han Chinese patients with type 2 diabetes will be recruited into the study through the Department of Endocrinology, Nanjing first Hospital. Following enrolment, patients will receive either an intensive insulin pump therapy for a months, or a combination of oral glucose-lowering agents (including metformin, DPP-4 inhibitors and/or sodium-glucose co-transporter-2 inhibitors), or a combination of oral glucose-lowering agents and injectable glucagon-like peptide-1 (GLP-1) receptor agonists for 3 months. Before the commencement of the therapy and on days 30 and 90, patients will attend the hospital for continuous glucose monitoring over 24 hours and measurement of gastric emptying using a 75 g oral glucose tolerance test (OGTT).

During their hospital stay, patients will consume 3 standard meals (i.e. breakfast, lunch and dinner) provided by the Department of Clinical Nutrition, with their glucose levels tracked by continuous glucose monitoring system (CGMS). Following the dinner, subjects will be asked to fast from solids and liquids (other than water) until the following morning, when they will be subjected to an OGTT at ~0900h. An intravenous cannula will be placed into a vein on the forearm. Subjects will be asked to consume a glucose drink containing 75 g glucose and 150mg 13C-acetate, within 5 min for the assessment of gastric emptying, postprandial glycemic and hormonal responses. Breath samples will be collected immediately before, and every 15 minutes after the drink for 3 hours for the measurement of gastric emptying. Venous blood samples will be taken at t = 0, 30, 60, 90, 120, 150 and 180 min for the measurements of plasma glucose, serum insulin, C-peptide, glucagon, total GLP-1, GIP and bile acids concentrations. Blood pressure and heart rate will be measured before and every 15 min after the drink for 3 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Patients newly diagnosed of type 2 diabetes as defined by published Criteria of World Health Organization in 1999; with HbA1c ≥ 7%, age ≥ 18 years of age and ≤ 80 years old, and willing to receive anti-diabetic treatments,
2. Non-diabetic controls, with BMI and age matched to patients with type 2 diabetes

Exclusion Criteria:

1. Patients with a fasting blood glucose ≤ 3.9mmol/L;
2. Patients with insulin allergy;
3. Patients with severe gastrointestinal symptoms and diseases;
4. Patients with gastrointestinal surgery history;
5. Use of any medication that may influence gastrointestinal motor function, body weight or appetite (opiates, anticholinergics, levodopa, clonidine, nitrates, tricyclic antidepressants, selective serotonin re-uptake inhibitors, phosphodiesterase type 5 inhibitors, sumatriptan, metoclopramide, domperidone, cisapride, prucalopride, or erythromycin);
6. Patients with major cardiovascular disease event (e.g., stroke, symptomatic peripheral artery disease, myocardial infarction, percutaneous coronary or peripheral artery angioplasty or coronary artery bypass surgery) in the previous 6 months;
7. Patients with liver dysfunction (aspartate aminotransferase or alanine aminotransferase level of more than two times the upper limit of normal range) or renal dysfunction (creatinine > 150 μmol/L or GFR < 60 mL/min/1.73m2);
8. Patients with severe anemia and hemoglobin disorders (Hb < 60 g/L);
9. Patients with infected injection site or coagulation disorders;
10. Patients who are pregnant.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Han Chinese patients newly diagnosed type 2 diabetes Han Chinese non-diabetic subjects
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2021-01-24 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Gastric-half emptying time of the 75 g glucose drink | Baseline, 1 month and 3 months in diabetic group
  The Change in gastric-half emptying time (min) before and after the treatment
Gastric-half emptying time of the 75 g glucose drink | Baseline in both diabetic and non-diabetic group
  The difference in gastric-half emptying time (min) between subjects with and without type 2 diabetes

SECONDARY OUTCOMES:
The mean blood glucose level | Baseline, 1 month and 3 months in the diabetic group
  The mean blood glucose level (mmol/L) during the 24 hours continuous glucose monitoring.
The mean amplitude of glycemic excursion | Baseline, 1 month and 3 months in the diabetic group
  The mean amplitude of glycemic excursion (mmol/L) during the 24 hours continuous glucose monitoring.
The percentage of blood glucose levels within the target range | Baseline, 1 month and 3 months in the diabetic group
  The percentage of blood glucose levels within the target range (%) during the 24 hours continuous glucose monitoring.
Serum insulin concentrations | t = 0, 30, 60, 120 and 180 min (t = 0 is when 75 g glucose drink is given) on baseline, 1 month and 3 months in the diabetic group
  The differences in the incremental under the curve from 0 to 180 min (iAUC0-180min) for serum insulin (mU/L) in response to a 75 g glucose drink before and after the treatment.
  The incremental area under the curve (iAUC) is calculated using the trapezoidal rule.
Serum C-peptide concentrations | t = 0, 30, 60, 120 and 180 min (t = 0 is when 75 g glucose drink is given) on baseline, 1 month and 3 months in the diabetic group
  The differences in the incremental area under the curve from 0 to 180 min (iAUC0-180min) for serum C-peptide (ng/mL) in response to a 75 g glucose drink before and after the treatment.
Serum total GLP-1 concentrations | t = 0, 30, 60, 120 and 180 min (t = 0 is when 75 g glucose drink is given) on baseline, 1 month and 3 months in the diabetic group
  The differences in the incremental under the curve from 0 to 180 min (iAUC0-180min) for serum total GLP-1 (pmol/L) in response to a 75 g glucose drink before and after the treatment.
Serum total GIP concentrations | t = 0, 30, 60, 120 and 180 min (t = 0 is when 75 g glucose drink is given) on baseline, 1 month and 3 months in the diabetic group
  The differences in the incremental under the curve from 0 to 180 min (iAUC0-180min) for serum total GIP (pmol/L) in response to a 75 g glucose drink before and after the treatment.
Serum bile acid concentrations | Baseline, 1 month and 3 months in the diabetic group
  The differences in the fasting serum bile acid concentrations (μmol/L) before and after the treatment.
Systolic blood pressure | t = 0, 15, 30, 45, 60,75, 90, 105, 120, 135, 150, 165 and 180 min (t = 0 is when 75 g glucose drink is given) on baseline, 1 month and 3 months in the diabetic group
  The differences in systolic blood pressure (mmHg) in response to the 75 g glucose drink before and after the treatment.
Diastolic blood pressure | t = 0, 15, 30, 45, 60,75, 90, 105, 120, 135, 150, 165 and 180 min (t = 0 is when 75 g glucose drink is given) on baseline, 1 month and 3 months in the diabetic group
  The differences in diastolic blood pressure (mmHg) in response to the 75 g glucose drink before and after the treatment.
Heart rate | t = 0, 15, 30, 45, 60,75, 90, 105, 120, 135, 150, 165 and 180 min (t = 0 is when 75 g glucose drink is given) on baseline, 1 month and 3 months in the diabetic group
  The differences in heart rate (beats/min) in response to the 75 g glucose drink before and after the treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Tongzhi Wu, PhD, Principal Investigator — The University of Adelaide; Jianhua Ma, PhD, Principal Investigator — The First Affiliated Hospital with Nanjing Medical University
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No
The ethical statement and informed consent do not allow for free data availability.

REFERENCES:
- [Background] Xie C, Huang W, Wang X, Trahair LG, Pham HT, Marathe CS, Young RL, Jones KL, Horowitz M, Rayner CK, Wu T. Gastric emptying in health and type 2 diabetes: An evaluation using a 75 g oral glucose drink. Diabetes Res Clin Pract. 2021 Jan;171:108610. doi: 10.1016/j.diabres.2020.108610. Epub 2020 Dec 7. PMID 33301790
- [Background] Wang X, Xie C, Marathe CS, Malbert CH, Horowitz M, Jones KL, Rayner CK, Sun Z, Wu T. Disparities in gastric emptying and postprandial glycaemia between Han Chinese and Caucasians with type 2 diabetes. Diabetes Res Clin Pract. 2020 Jan;159:107951. doi: 10.1016/j.diabres.2019.107951. Epub 2019 Nov 29. PMID 31790715
- [Background] Goyal RK. Gastric Emptying Abnormalities in Diabetes Mellitus. N Engl J Med. 2021 May 6;384(18):1742-1751. doi: 10.1056/NEJMra2020927. No abstract available. PMID 33951363
- [Background] Watson LE, Xie C, Wang X, Li Z, Phillips LK, Sun Z, Jones KL, Horowitz M, Rayner CK, Wu T. Gastric Emptying in Patients With Well-Controlled Type 2 Diabetes Compared With Young and Older Control Subjects Without Diabetes. J Clin Endocrinol Metab. 2019 Aug 1;104(8):3311-3319. doi: 10.1210/jc.2018-02736. PMID 30933282
- [Background] Phillips LK, Deane AM, Jones KL, Rayner CK, Horowitz M. Gastric emptying and glycaemia in health and diabetes mellitus. Nat Rev Endocrinol. 2015 Feb;11(2):112-28. doi: 10.1038/nrendo.2014.202. Epub 2014 Nov 25. PMID 25421372